CLINICAL TRIAL: NCT01715441
Title: A Randomized Phase II Trial Assessing Sorafenib in Combination With Irinotecan in Metastatic Colorectal Cancer Patients With KRAS Mutated Tumors After Failure of All Drugs Known to be Effective
Brief Title: Sorafenib in Combination With Irinotecan in Metastatic Colorectal Cancer Patients With KRAS Mutated Tumors
Acronym: NEXIRI2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEXIRI2; 2012-000644-94 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-29 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer Patients With KRAS Mutated Tumors
Keywords: Metastatic colorectal cancer patients; KRAS mutation; Sorafenib
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Irinotecan monotherapy (Active Comparator): Intravenous infusion irinotecan 180 mg/m2 over 90 minutes (D1=D15) with cross over to irinotecan and sorafenib combination at progression.
  Interventions: Drug: Irinotecan monotherapy
- Sorafenib monotherapy (Active Comparator): Oral sorafenib 400 mg twice daily (total dose 800 mg/day) with cross over to irinotecan and sorafenib combination at progression
  Interventions: Drug: Sorafenib monotherapy
- Sorafenib and irinotecan combination (Experimental): Intravenous infusion irinotecan 120 mg/m2 over 90 minutes (D1=D15) at Cycle 1, 150 mg/m² at C2 if no diarrhea > grade 1 and no other toxicity > grade 2, and 180 mg/m² at C3 in the same conditions
  * Oral sorafenib 400 mg twice daily (total dose 800 mg/day) from C1. 1 cycle = 15 days and 1 course = 4 weeks.
  Interventions: Drug: Sorafenib and irinotecan combination

INTERVENTIONS:
Drug: Sorafenib and irinotecan combination
  Arms: Sorafenib and irinotecan combination
Drug: Sorafenib monotherapy
  Arms: Sorafenib monotherapy
Drug: Irinotecan monotherapy
  Arms: Irinotecan monotherapy

SUMMARY:
The aim of this multicenter randomized phase II trial is to determine the efficacy of sorafenib and irinotecan combination versus irinotecan monotherapy or versus sorafenib monotherapy in metastatic colorectal cancer patients with KRAS mutated tumors after failure of all active drugs known to be effective.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* Histologically confirmed diagnosis of colorectal cancer
* Asymptomatic or resected primary tumor
* Metastatic colorectal cancer patient not eligible for curative surgery
* At least one target lesion:

  * Unidimensionally measurable on cross-sectional imaging
  * In an area not previously irradiated
* Disease progression after failure of active drugs (5-Fu or 5-Fu prodrugs, irinotecan, oxaliplatin, bevacizumab)
* Patients with bone metastases are eligible if they have other measurable lesions
* WHO performance status ≤ 2
* Confirmation of KRAS mutation in codons 12 or 13 in the primary tumor or metastases
* Total bilirubin ≤ 1.5 ULN, ALT or AST ≤ 2.5 ULN (or < 5 in case of liver impairment)
* Haemoglobin ≥ 10 g/dL, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3
* Serum creatinine ≤ 1.5 ULN
* Negative pregnancy test in women of childbearing potential
* Use of an effective contraceptive method during the whole treatment and up to 3 months after the completion of treatment in males and females
* Life expectancy of at least 3 months
* Informed consent signed prior any study specific procedures
* Tumor evaluation should be performed within 3 weeks prior to starting treatment

Exclusion Criteria:

* History of Gilbert's syndrome
* Symptomatic brain metastases or carcinomatous meningitis
* Bone-only metastases
* History or presence of other cancers within the past 5 years (except curatively treated non-melanoma skin cancer and in situ cervical cancer)
* Prior surgery or radiotherapy within 4 weeks before entering the study
* Cardiac arrhythmia requiring treatment (except for beta-blockers and digoxin), unstable cardiac disease, myocardial infarction within the previous 6 months, > grade II NYHA heart failure, uncontrolled hypertension
* Kalemia lower than normal serum potassium value
* From ECG, QTc interval > 470 ms
* History of acute or chronic pancreatitis
* History of epileptic seizures requiring long-term anticonvulsant therapy
* History of organ transplantation with use of immunosuppression therapy
* Severe bacterial or fungal infection (Grade > 2 NCI-CTCAE v.4.0)
* Known HIV infection
* Long-term use of CYP 3A4 enzyme-inducing agents such as rifampicin, St. John's Wort (hypericum perforatum), phenytoin, carbamazepine, phenobarbital, dexamethasone, and ketoconazole
* Pregnant or breastfeeding women
* Bowel malabsorption or extended bowel resection that could affect the absorption of sorafenib, occlusive syndrome, inability to take oral medications
* Inflammatory bowel disease with chronic diarrhea (NCI-CTCAE v.4.0)
* Participation in another clinical trial 30 days prior to study entry
* Concurrent treatment with any other investigational product or anticancer therapy (except for irinotecan or sorafenib)
* Psychological, social, geographical disorders or any other condition that would preclude study compliance (treatment administration and study follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Non-progression rate | At 2 months
  To evaluate the non-progression rate at 2 months according to RECIST criteria (Version 1.1)

SECONDARY OUTCOMES:
Disease control rate | At 2 months
  According to RECIST criteria (Version 1.1)
Treatment-related toxicity | At 6 months
  According to NCI CTC V4.0
Overall survival | At 6 months
  Overall survival is defined as the time from the date of inclusion to the date of death from any cause.
Quality of life questionnaire | 6 months
  Using the EORTC QLQ-C30 questionnaire
Progression Free Survival | At 6 months
  Progression Free Survival is defined as the time from the date of inclusion to first documentation of objective tumor progression or to death due to progression.
Response rate | At 2 months
  According to RECIST criteria (Version 1.1)

OTHER OUTCOMES:
Cmax and Tmax of sorafenib and irinotecan | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle SAMALIN, MD, Principal Investigator — CRLC Val d'Aurelle-Paul Lamarque; Marc YCHOU, MD,, Study Chair — CRLC Val d'Aurelle
Locations (9):
- France (9):
  - Hôpital AVICENNE, Bobigny
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital LA TIMONE, Marseille
  - CRLC Val d'Aurelle-Paul Lamarque, Montpellier
  - C.H.U. de REIMS, Reims
  - CHU Charles Nicolle, Rouen
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain

REFERENCES:
- [Result] Samalin E, Fouchardiere C, Thezenas S, Boige V, Senellart H, Guimbaud R, Taieb J, Francois E, Galais MP, Lievre A, Seitz JF, Metges JP, Bouche O, Boissiere-Michot F, Lopez-Crapez E, Bibeau F, Ho-Pun-Cheung A, Ychou M, Adenis A, Di Fiore F, Mazard T. Sorafenib Plus Irinotecan Combination in Patients With RAS-mutated Metastatic Colorectal Cancer Refractory To Standard Combined Chemotherapies: A Multicenter, Randomized Phase 2 Trial (NEXIRI-2/PRODIGE 27). Clin Colorectal Cancer. 2020 Dec;19(4):301-310.e1. doi: 10.1016/j.clcc.2020.04.008. Epub 2020 May 15. PMID 32737004